CLINICAL TRIAL: NCT04124822
Title: Effectiveness of Single Dose Pre Medication of Piroxicam and Prednisolone on Post Endodontic Pain After a One Visit Root Canal Treatment. Randomized Trial .
Brief Title: Effectiveness if Premedication With Single Dose Piroxicam and Prednisolone After a Single Visit Root Canal Treatment .
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Anum Tanwir , MDS, MDS trainee (operative dentistry), Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dikiohs2013
Record Dates: First submitted 2019-08-19; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Post-operative Endodontic Pain
MeSH Terms: interventions — Piroxicam; Prednisolone

STUDY DESIGN:
Intervention Model Description: subjects are randomly placed into one of the three groups: Placebo, Piroxicam (20 mg), Prednisolone (20 mg). The drugs will be given thirty minutes before procedure starts,followed by one visit root canal procedure. Postoperative pain will be evaluated up to 96 hours interval using a visual analog scale.
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is a double blinded study in which investigator /caregiver and participant will be blinded and 3rd person not in the study will be dispatching drugs from the coded bottles .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (No Intervention): group 1 , is no intervention group in which root canal procedure will be done without drug as ideal protocol .
- Piroxicam (Experimental): group 2 is given Piroxicam 20 mg half an hour before root canal treatment to manage post operative pain.
  Interventions: Drug: Piroxicam 20 mg
- Prednisolone (Experimental): group 3 is given Prednisolone 20mg half an hour before root canal treatment to manage post operative pain.
  Interventions: Drug: prednisolone 20 mg

INTERVENTIONS:
Drug: Piroxicam 20 mg — Piroxicm is from oxicam family of anti inflammatory drug that inhibits prostaglandin synthesis and effectively lower pain threshold levels
  Arms: Piroxicam
Drug: prednisolone 20 mg — prednisolone is from steroid family of anti inflammatory drug that inhibit arachidonic acid and effectively lowers the pain
  Arms: Prednisolone

SUMMARY:
Two drugs (Piroxicam and Prednisolone)are being compared for post operative endodontic pain after a single visit root canal treatment for 74 hours.

DETAILED DESCRIPTION:
To evaluate effectiveness of single dose premedication with piroxicam(20mg) and prednisolone(20mg) on post endodontic pain after a single visit root canal treatment .

patient will be recalled every day for 4 days to know the pain scale using visual analogue scale .

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages from 20-40 years(28).
2. Single rooted tooth with symptomatic irreversible pulpitis.
3. With no analgesic or anti-inflammatory drug taken within a week period before procedure.

Exclusion Criteria:

1. Patients presenting with any systemic disease
2. Patients already taking premedication for endodontic pain.
3. Pregnant or lactating patients.
4. Multirooted teeth.
5. Teeth with Pulpal necrosis.
6. Previously treated or initiated root canal treatment.
7. Patient presenting with allergy due to drug

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
post operative pain | 76 hours
  post operative pain will be measured after single visit endodontic treatment using visual analog scale with readings 1 to 10 from 24 hours till 76 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anum Tanwir, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- DUHS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanwir A, Ahmed S, Akhtar H, Wahid U, Shakoor Abbasi M, Ahmed N. Effectiveness of Single Dose Premedication of Piroxicam and Prednisolone on Post Endodontic Pain in One Visit Root Canal Treatment: A Randomized Clinical Trial. Eur Endod J. 2022 Oct;7(3):187-192. doi: 10.14744/eej.2022.24119. PMID 36217645